CLINICAL TRIAL: NCT07362862
Title: Safety and Feasibility of the MyokinE100 System in ICU Settings to Mitigate ICU Acquired Weakness
Brief Title: MyokinE100 System: Closed Loop Electrical Muscle Stimulation to Mitigate ICU Acquired Weakness in Medical ICU Patients
Acronym: ICUAW
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Health Discovery Labs (Industry)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH); Mayo Clinic (Other); Ascension Health (Industry); University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00006725; R44EB033725 (NIH)
Record Dates: First submitted 2025-12-19; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Sepsis; Critical Illness; ICU-acquired Muscle Weakness; ICU-acquired Weakness; ICUAW; Sarcopenia; Secondary Sarcopenia
Keywords: Electrical muscle stimulation; Electrical Impedance Myography; Bioimpedance; Rehabilitation; Sepsis; Critical illness; ICU-acquired weakness
MeSH Terms: conditions — Sepsis; Critical Illness; Sarcopenia

STUDY DESIGN:
Intervention Model Description: Two groups of participants will each receive different interventions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Intervention Group (Active Comparator): Participants will receive a daily 60-minute session of electrical muscle stimulation applied to the quadriceps for up to 7 days during ICU stay or until ICU discharge, alongside standard of care.
  Interventions: Device: Electrical Muscle Stimulation System
- Control Group (No Intervention): Participants will receive standard of care only

INTERVENTIONS:
Device: Electrical Muscle Stimulation System — Participants will receive electrical muscle stimulation at the level of the quadriceps using the MyokinE100 device, a closed-loop electrical muscle stimulation system.
  The closed-loop system monitors muscle response to electrical stimulation in real time using a biofeedback sensor and automatically adjusts stimulation intensity to achieve safe and effective muscle contractions.
  Arms: Intervention Group

SUMMARY:
The goal of this clinical trial is to learn if a new medical device that sends electrical signals to the thigh muscles is safe and easy to use for people in the ICU (Intensive Care Unit) who are at risk of losing muscle strength. It will also explore whether this treatment can help slow down muscle weakening.

The main questions this study aims to answer are:

* Do participants develop medical problems when receiving electrical muscle stimulation in the ICU?
* Is electrical muscle stimulation a practical way to help reduce muscle weakness in critically ill patients?

Researchers will compare the control group (standard of care) to the intervention group (standard of care plus 60-minute sessions of electrical muscle stimulation daily during the ICU stay) to see if the device is safe and easy to use.

Participants will:

* Receive either standard of care or standard of care plus electrical muscle stimulation of the thigh muscles
* Have their muscle strength checked during the study
* Complete a survey three months after ICU discharge to check on their recovery

ELIGIBILITY:
Inclusion Criteria:

* Admitted to ER or ICU within the previous 48 hours
* APACHE II score ≥ 13
* Meets the criteria for sepsis or severe sepsis
* Baseline Clinical Frailty Scale (CFS) ≤ 4

Exclusion Criteria:

* Anticipated transfer to an ICU not participating in this study
* Expected length of ICU stay < 48 hours
* Myopathies (e.g. congenital)
* Acquired myopathies with CK levels 5-times above the upper limit of normal
* Unable to transfer from bed to chair at baseline
* Moribund
* Comfort care
* New onset deep vein thrombosis within the previous 6-months
* Malignancy in lower limb
* Technical obstacles - fracture, burns, amputation
* Open wound or skin abrasion at the garment application site
* Pregnancy
* Pacemaker and implantable cardioverter-defibrillator

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in lower limb muscle strength assessed by MRC sum score from ICU admission to ICU discharge. | Day 1 (day of enrollment) and daily in the ICU up to Day 14 or upon ICU discharge whichever comes first.
  Lower limb muscle strength will be assessed using the Medical Research Council (MRC) sum score. The MRC sum score grades voluntary muscle contraction for each muscle group from 0 (no contraction) to 5 (normal strength). Six muscle groups in lower limbs will be tested for a total best possible score of 30.
  A 1-point increase in MRC score per muscle group in the lower limbs is considered clinically significant.
Number of participants with unanticipated adverse device effects (UADE) related to MyokinE100 use from enrollment to hospital discharge. | From Day 1 (enrollment) through the end of the subject's study participation at 3-months.
  A single Unanticipated Adverse Device Effect (UADE) in any participant during the study is considered significant.

SECONDARY OUTCOMES:
Change in total muscle strength assessed by MRC sum score from ICU admission to ICU discharge. | Day 1 (day of enrollment) and daily in the ICU up to Day 14 or upon ICU discharge whichever comes first.
  Upper and lower limb muscle strength will be assessed using the Medical Research Council (MRC) sum score. The MRC sum score scale grades voluntary muscle contraction for each muscle group from 0 (no contraction) to 5 (normal strength). Twelve muscle groups will be tested for a total possible best score of 60.
  A 1-point change in MRC sum score is considered clinically significant.
Change in hand-grip muscle strength measured by handheld dynamometry from ICU admission to hospital discharge. | Day 1 (day of enrollment) and daily in the ICU up to Day 14, and on hospital discharge day.
  Handgrip muscle strength will be assessed using a handheld dynamometer (HHD) as an indicator of global muscle function. Participants will be considered to have ICU-Acquired Weakness (ICUAW) if the average handgrip strength is below the threshold of 11Kg for men or 7 Kg for woman.
  Higher scores in Kg indicate greater global muscle function.
Change in mobility status assessed by ICU Mobility Scale (IMS) from ICU admission to ICU discharge. | Day 1 (day of enrollment) and daily in the ICU up to Day 14 or upon ICU discharge whichever comes first.
  Functional mobility will be assessed using the ICU Mobility Scale (IMS), which ranges from 0 (lying in bed, no active movement) to 10 (walking independently without a gait aid).
  Higher scores indicate greater mobility.
Change in functional exercise capacity assessed by Six-Minute Walk Test (6MWT) between ICU discharge to hospital discharge. | Measured on the day of ICU discharge, average day 7, and on the day of hospital discharge, average day 14.
  Functional exercise capacity will be assessed using the Six-Minute Walk Test (6MWT) which measures the distance a participant can walk on a flat surface in six minutes.
  A greater distance walked indicates better functional status.
Change in functional exercise capacity assessed by 30-Second Sit-to-Stand Test (30 s STS) between ICU discharge to hospital discharge. | Measured on the day of ICU discharge, average day 7, and on the day of hospital discharge, average day 14.
  Functional exercise capacity will be assessed using the 30-Second Sit-to-Stand Test (30 s STS) which measures how many times a person can stand up from and sit down (one repetition) in an armless chair in 30 seconds.
  A higher number of repetitions indicates greater functional capacity.
Change in Rectus Femoris muscle structure assessed by musculoskeletal ultrasound from ICU admission to hospital discharge. | From ICU admission to day 14.
  The Rectus Femoris muscle structure will be evaluated using musculoskeletal ultrasound. Measurements will include cross-sectional area, muscle circumference, pennation angle, and echo-intensity.
  Higher cross-sectional area, muscle circumference, and pennation angle indicate better muscle structure, while increased echo-intensity suggests worse muscle structure.
Change in frailty status assessed by Clinical Frailty Scale (CFS) from ICU admission to 3-month post hospital discharge. | Enrollment to 3-month follow-up.
  Frailty will be assessed using the Clinical Frailty Scale (CFS), which ranges from 1 (very fit) to 7 (severely frail).
  Higher scores are worse.
Change in functional independence assessed by Barthel Index from ICU discharge to hospital discharge. | Enrollment to 3-month follow-up.
  Functional independence will be assessed using the Barthel Index, which measures patient's ability in 10 activities of daily living (feeding, bathing, grooming, dressing, bowel control, bladder control, toilet use, chair transfers, mobility on level surfaces, and stairs).
  A higher score closer to 100 indicate greater functional independence.
Change in fatigue severity assessed by Visual Analog Scale for Fatigue (VAS-F) from ICU admission to hospital discharge. | From ICU admission up to Day 14 or upon ICU discharge whichever comes first.
  Fatigue will be assessed using the Visual Analog Scale for Fatigue (VAS-F), where participants rate their fatigue on a scale from 0 (no fatigue) to 10 (worst possible fatigue).
  Higher scores indicate greater fatigue.
Change in health-related quality of life assessed by the RAND 36-Item Health Survey (SF-36) from the time of hospital discharge to 3-month follow-up after hospital discharge. | Hospital discharge to 3-month follow-up after hospital discharge.
  Health-related quality of life will be assessed using the RAND 36-Item Health Survey (SF-36), which evaluates eight domains including physical functioning, role limitations, pain, general health, vitality, social functioning, emotional well-being, and mental health. Scores range from 0 to 100, with higher scores indicating better health status.
Change in employment status and work ability after hospital discharge. | From ICU discharge to 3-month follow up after hospital discharge.
  Employment status will be assessed during follow-up after hospital discharge using a structured questionnaire. Participants will report their current employment status and whether their ICU stay affected their ability to work.
  Return to work is considered best outcome.
Duration of mechanical ventilation. | From ICU admission to ICU discharge, an average of 7 days.
  The number of days from the initiation of mechanical ventilation to the discontinuation of mechanical ventilation.
  A lower number of days is better.
Number of ventilator-free days within 28 days after ICU admission. | From extubation to day 28.
  Ventilator-free days will be calculated as 28 minus total number of days on invasive mechanical ventilation during which the participant is alive and not receiving invasive mechanical ventilation.
  Participants who die within 28 days will be assigned zero ventilator-free days.
Number of days in ICU, hospital ward, and total hospital stay from admission to discharge. | From hospital admission to hospital discharge, an average of 14 days.
  Length of stay will be recorded in three categories: (1) ICU stay, defined as the total number of consecutive days from ICU admission to ICU discharge; (2) ward stay, defined as the number of days spent in a hospital ward after ICU discharge; and (3) total hospital stay, defined as the number of days from hospital admission to hospital discharge.
  The shorter the length of stay, the better.
Discharge location after hospital stay. | At the last day of hospitalization, average day 14.
  Discharge location will be recorded at the time of hospital discharge using predefined categories: home, home with home health services, inpatient rehabilitation facility, skilled nursing facility, long-term acute care hospital, hospice, or death.
  Discharge home is considered the best outcome.
Number of participants tolerating electrical muscle stimulation sessions during ICU stay. | From day 1 in the ICU up to 7 days or ICU discharge whichever comes first.
  Treatment session tolerance will be assessed using standardized scales.
  Tolerance is defined as:
  * CPOT less than 7
  * NRS less than 8 at the thigh level
  * RASS less than +3
  Scale ranges:
  * CPOT (0 = relaxed, 8 = severe pain/agitation)
  * NRS for pain (0 = no pain, 10 = worst pain),
  * RASS (-5 = unarousable, +4 = combative)
Number of participants with electrical interference on ECG monitoring during the stimulation sessions in the ICU. | From day 1 in the ICU up to 7 days or ICU discharge whichever comes first.
  Electrical interference with cardiac monitoring will be assessed during each electrical muscle stimulation (EMS) session using ECG tracings from standard ICU cardiac monitoring devices. Interference is defined as continuous 60-cycle (60 Hz) artifact for more than 60 seconds that impairs accurate interpretation of cardiac rhythm. ECG data will be captured only during EMS intervention sessions.
  Success is defined as 20% or less of ECG samples showing electrical interference as defined above.
Number of participants achieving significant muscle contraction during electrical muscle stimulation sessions as assessed by Muscle Contraction Scale during the ICU stay. | From day 1 in the ICU up to 7 days or ICU discharge whichever comes first.
  "Muscle contraction during electrical muscle stimulation (EMS) sessions will be assessed using the Muscle Contraction Scale, which classifies contraction from Type 1 (no palpable or visible contraction) to Type 5 (palpable and visible contraction with full muscle bulk).
  Participants achieved a response if they scored muscle contraction grade 3 or higher.

OTHER OUTCOMES:
Change in Impedance (Z), Reactance (X), and Phase Angle (PA) of the quadriceps muscle during the hospital stay. | From day 1 up to hospital discharge or day 14 whichever comes first.
  Quadriceps muscle electrical properties will be measured using Electrical Impedance Myography (EIM). Measurements will include Impedance (Z in ohms), Reactance (X in ohms), and Phase Angle (PA in degrees), which reflect muscle composition.
  Lower Phase Angle and Reactance values indicate reduced muscle composition. Higher Impedance values generally indicate reduced muscle health.
Change in C-Terminal Agrin Fragment (CAF) level in blood and urine from enrollment to day 14. | From enrollment to day 14.
  C-Terminal Agrin Fragment (CAF) levels will be measured in blood and urine samples collected from enrollment through Day 14. Higher CAF levels may indicate increased neuromuscular junction degradation, while lower levels suggest better preservation of muscle function.

CONTACTS AND LOCATIONS:
Overall Officials: Oussama Hassan, M.D., Principal Investigator — Health Discovery Labs
Locations (3):
- United States (3):
  - Mayo Clinic, Rochester, Minnesota
  - Dell Seton Medical Center at The University of Texas, Austin, Texas
  - Ascension Seton Medical Center Austin, Austin, Texas

IPD SHARING:
Plan to Share IPD: Undecided